CLINICAL TRIAL: NCT03318679
Title: "Is Non Diabetic Hyperglycemia in Acute Ischemic Stroke Part of a Systemic Stress Response"
Brief Title: Assessment of Markers of Stress in Acute Ischemic Stroke With Hyperglycemia
Acronym: ASIIST
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: UMinnesota
Record Dates: First submitted 2017-09-25; First posted 2017-10-24 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Ischemic Stroke; Hyperglycemia
MeSH Terms: conditions — Ischemic Stroke; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention is planned. — None is planned

SUMMARY:
Hyperglycemia is present in 50 percent of patients with acute ischemic stroke. Patients with hyperglycemia have higher in hospital, 30 and 90 day mortality and morbidity. Sixty percent of these patients have some form of diabetic syndrome, known or unknown. Remaining 40% of patients are not diabetic. Contrary to logic patients with non diabetic hyperglycemia (NDH) have statistically higher morbidity and mortality compared to the diabetic hyperglycemia (DH) cohort. So far multiple treatment trials (THIS, GRASP, GIST-UK, SHINE ongoing) with differing treatment goals have shown no clear benefit, however no obvious distinction was made along the diabetic and non-diabetic hyperglycemic groups.

If hyperglycemia in the acute phase was the only culprit in worsening the injury, then there should be no difference in the outcomes for DH and NDH. Existing data implies that the two categories are two distinct physiological entities that are thus not amenable to same treatment. Stating it simply NDH is not an insulin deficient state where as DH is.

Alternative possibility is that body and Neurons are accustomed to high sugars in diabetics and thus can tolerate higher sugars better during ischemic stroke compared to non diabetics.

The overarching hypothesis is that reducing blood sugars in NDH increases stroke volume and thus consequently worsens outcome.

DETAILED DESCRIPTION:
1.1 Background Hyperglycemia is present in 50 percent of patients with acute ischemic stroke. Patients with hyperglycemia have higher in hospital, 30 and 90 day mortality and morbidity. Sixty percent of these patients have some form of diabetic syndrome, known or unknown. Remaining 40% of patients are not diabetic. Contrary to logic patients with non diabetic hyperglycemia (NDH) have statistically higher morbidity and mortality compared to the diabetic hyperglycemia (DH) cohort. So far multiple treatment trials (THIS, GRASP, GIST-UK, SHINE ongoing) with different treatment goals have shown no clear benefit.

If hyperglycemia in the acute phase was the only culprit in worsening the injury, then there should be no difference in the outcomes for DH and NDH. Existing data implies that the two categories are distinct physiological entities that are thus not amenable to same treatment. Stating it simply NDH is not an insulin deficient state where as DH is.

Alternative possibility is that body and Neurons are accustomed to high sugars in diabetics and thus can tolerate higher sugars better during ischemic stroke compared to non diabetics.

The overarching hypothesis is that reducing blood sugars in NDH increases stroke volume and thus consequently worsens outcome.

1.2 Investigational Agent: No planned investigational agent is tested as part of this study.

1.3 Pre-clinical Data Currently there is clear data that patients that present with acute ischemic stroke have higher (two times) mortality at discharge and 90 day mark. Multiple clinical studies so far have not revealed any clear benefit of treatment (GIST-UK). There do seem to be two distinct groups when it comes to hyperglycemia at presentation of DM, HG in association of Diabetes and without any history of Diabetes. The outcomes in the two groups vary greatly.

1.4 Clinical Data to Date Please see attached article with references.

1.5 Dose Rationale and Risk/Benefits There is no drug or device or intervention that will be tested in this study. This study involves collection of blood samples from the patients who meet the inclusion criteria. Our goal is to be able to see if there is any difference between the two groups of patients.

2 Study Objectives

Primary Objective: Assess difference in laboratory values between two groups of patients.

Null Hypothesis: There is no difference in laboratory values between DH and NDH

3 Study Design

3.1 General Design This is a exploratory study to assess the difference in the lab values in two groups of patients. Patients that present to University of Minnesota Medical Center with acute ischemic stroke and are hyperglycemic (Blood sugar of more than 130 mg/dl) will be eligible for the study. Pre-specified volume of blood will be collected for lab analysis. This study does not involve testing of any procedure, drug or device.

Step One - Identify patients that have Ischemic strokes and have hyperglycemia >130 mg/dl.

Step Two:

- Obtain Consent from patient or POA.

Step Three:(Once consent obtained) - Collect first set of blood samples from patients with the first blood draw between 0-8 hours from time of ER arrival. Second blood sample will be collected in 9-16 hours and a 3rd one in 17-24 hour period.

Step Four:

- No further data will be collected from patient. Study end point is difference in laboratory values between DH and NDH groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute Ischemic stroke that present to UMMC ER.
2. Age 18-100.
3. Subjects are hyperglycemic (defined as blood sugar above 130mg/dl).

Exclusion Criteria:

1. Blood sugars less than 130mg/dl.
2. Age less than 18 or more than 100.
3. Difficult blood draw.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acute Ischemic Stroke Patients that present to University of Minnesota Medical Center and Hennipen County medical Center.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Difference in the Bio markers of stress between Diabetic and Non diabetic patients that have acute ischemic stroke and hyperglycemia on presentation. | 24 hours
  Lab values

CONTACTS AND LOCATIONS:
Overall Officials: Rwoof A Reshi, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reshi R, Streib C, Ezzeddine M, Biros M, Miller B, Lakshminarayan K, Anderson D, Ardelt A. Hyperglycemia in acute ischemic stroke: Is it time to re-evaluate our understanding? Med Hypotheses. 2017 Sep;107:78-80. doi: 10.1016/j.mehy.2017.08.017. Epub 2017 Aug 16. PMID 28915969
- See also: Hyperglycemia in acute ischemic stroke: Is it time to re-evaluate our understanding? — https://www.ncbi.nlm.nih.gov/pubmed/28915969